CLINICAL TRIAL: NCT05300282
Title: A Phase I/II b (Randomized Controlled) Study of Atezolizumab Combined to BEGEV Regimen as First Salvage Treatment in Patients With Relapsed or Refractory Hodgkin's Lymphoma Candidate to Autologous Stem-Cell Transplantation
Brief Title: Study of Atezolizumab Plus BEGEV Regimen in Relapsed or Refractory Hodgkin's Lymphoma Patients
Acronym: FIL_A-BEGEV
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FIL_A-BEGEV
Record Dates: First submitted 2022-03-08; First posted 2022-03-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Relapsed or Refractory Hodgkin's Lymphoma
Keywords: Hodgkin's lymphoma; atezolizumab; BEGEV; phase I/II b study; relapsed; refractory; MTD
MeSH Terms: conditions — Recurrence; Hodgkin Disease | interventions — atezolizumab; Bendamustine Hydrochloride; Gemcitabine; Vinorelbine

STUDY DESIGN:
Intervention Model Description: The phase I part is aimed at determining the MTD of atezolizumab when combined with BEGEV schedule. Atezolizumab dosing starts at 1200 mg and decreases in the successive cohort to the dose of 840 mg and 600 mg to reach MTD which will be used in the phase II part where patients will be randomized in 2 arms: arm A will receive the BEGEV regimen followed by ASCT for patients achieving CR and arm B will receive combination treatment with Atezolizumab and BEGEV regimen followed for patients reaching CR by ASCT plus a consolidation with 6 doses of atezolizumab at 1200 mg every 4 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- phase I (Experimental): patients will receive the BEGEV regimen plus Atezolizumab in order to determine MTD of the last one drug.
  Interventions: Drug: Atezolizumab; Combination Product: BEGEV
- phase IIb - arm A (Active Comparator): patients will receive the BEGEV regimen followed by ASCT for patients achieving CR.
  Interventions: Combination Product: BEGEV
- phase IIb - arm B (Experimental): patients will receive combination treatment with Atezolizumab (at dose obtained from phase I) and BEGEV regimen followed for patients reaching CR by ASCT plus a consolidation with 6 doses of atezolizumab at 1200 mg every 4 weeks.
  Interventions: Drug: Atezolizumab; Combination Product: BEGEV

INTERVENTIONS:
Drug: Atezolizumab — In phase I study: Atezolizumab will be administered until the determination of its MTD when combined with BEGEV schedule.
  In phase II b study - arm A (standard): Atezolizumab will not be administered. In phase II b study - arm B (experimental): Atezolizumab will be administered at MTD determined in phase I study plus BEGEV regimen (at dosages performed by local practice).
  Arms: phase I; phase IIb - arm B
Combination Product: BEGEV — In phase I study: Atezolizumab will be administered until the determination of its MTD when combined with BEGEV schedule.
  In phase II b study - arm A (standard): only BEGEV will be administered. In phase II b study - arm B (experimental): BEGEV regimen will be administered in combination with Atezolizumab at MTD determined in phase I.
  Other Names: Bendamustine; Gemcitabine; Vinorelbine

SUMMARY:
The phase I part (safety assessment of the combination treatment) is aimed at determining the MTD of atezolizumab when combined with BEGEV schedule.

6-18 patients enrolled in this part will be treated with atezolizumab in combination with BEGEV regimen every 3 weeks for 4 cycles.

Patients without a DLT in the first cycle and without disease progression after cycle 2, will undergo stem cell mobilization with 3-4 cycle of A-BEGEV + granulocyte colony-stimulating factor (G-CSF) and subsequently receive a myeloablative therapy followed by ASCT.

The phase IIb part (expansion cohort) plans to randomize 122 patients in two arms (A and B, 61 per arm):

1. arm A will receive the BEGEV regimen followed by ASCT for patients achieving CR.
2. arm B will receive combination treatment with Atezolizumab and BEGEV regimen followed for patients reaching CR by ASCT plus a consolidation with 6 doses of atezolizumab at 1200 mg every 4 weeks.

After the last treatment date of the last patient (LPLT), the phase IIb will be ended. A long term follow up will start, in order to better assess patients' prognosis. All evaluable patients from phase I and phase IIb study will enter in the long term follow up phase and will be followed for 18 months.

DETAILED DESCRIPTION:
The phase I part (safety assessment of the combination treatment) is aimed at determining the MTD of atezolizumab when combined with BEGEV schedule.

6-18 patients enrolled in this phase will be treated with atezolizumab in combination with BEGEV regimen every 3 weeks for 4 cycles.

Patients without a DLT in the first cycle and without disease progression after cycle 2, will undergo stem cell mobilization with 3-4 cycle of A-BEGEV + granulocyte colony-stimulating factor (G-CSF) and subsequently receive a myeloablative therapy followed by ASCT.

Patients with documented CR following ASCT will receive a consolidation therapy with atezolizumab as single agent every 4 weeks for 6 doses, starting preferably between 60 and 90 days, but ≥ 60 days and not > 120 days after autografting. In patients not previously radiotreated, adjuvant radiotherapy (RT) should be planned during consolidation treatment within the start of second consolidation dose, according to clinician's judgment and response assessment. RT will be administered at 30-36 Gy on sites of initial bulky disease or on single PET positive residual site.

Patients reaching PR after four cycles of atezolizumab combined with BEGEV or with documented PR after ASCT may continue the study protocol according to the physician judgment.

Dosing starts at 1200 mg and decreases in the successive cohort to the dose of 840 mg and 600 mg, according to Flow chart A. in the section 6 of the protocol.

In the consolidation phase atezolizumab will be administered at dose of 1200 mg every 4 weeks for 6 doses without dose reduction, but only delay or discontinuation.

Patients included in the cohort developing DLT, withdraw the protocol due to toxicity and continue the treatment according to good clinical practice.

For patients included in the cohort of MTD, monitoring and collection of AEs will be continuous during induction, consolidation treatment and follow-up.

The phase IIb part (expansion cohort) plans to randomize 122 patients in two arms (A and B, 61 per arm):

1. arm A will receive the BEGEV regimen followed by ASCT for patients achieving CR.
2. arm B will receive combination treatment with Atezolizumab and BEGEV regimen followed for patients reaching CR by ASCT plus a consolidation with 6 doses of atezolizumab at 1200 mg every 4 weeks.

In patients not previously radiotreated, adjuvant RT should be planned for both patients in arm A and arm B according to clinician's judgment and response assessment. RT will be administered at 30-36 Gy on sites of initial bulky disease or on single PET positive residual site.

Patients reaching PR after four induction cycles (atezolizumab combined with BEGEV or BEGEV alone) or with documented PR after ASCT may continue the study protocol according to the physician judgment.

After the last treatment date of the last patient (LPLT), the phase IIb will be ended. A long term follow up will start, in order to better assess patients' prognosis. All evaluable patients from phase I and phase IIb study will enter in the long term follow up phase and will be followed for 18 months. Disease status, survival outcome, secondary primary malignancies and late toxicity will be collected every 6 months until patient withdrawal of consent, lost to follow up and patient's death. Long term follow-up phase will end 18 months after the end of phase IIb.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old (upper limit valid only for phase I).
* Histologically confirmed cHL, at first disease relapse or refractory to a first-line treatment or with documented persistent disease at interim positron emission tomography (PET) performed after 2 cycles of first line (ABVD/ABVD like/BEACOPP).
* Only one prior systemic therapy for Hodgkin's lymphoma (HL).
* First disease relapse or refractory to a first-line treatment.
* Eligibility for ASCT.
* Performance status (PS) ≤ 2 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Adequate haematological function, unless abnormalities due to underlying disease, at the moment of signing informed consent, defined as follows:

  * neutrophils > or = 1.500/mmc and
  * platelets > or = 75.000/mmc and
  * haemoglobin > or = 8,0 g/dL with transfusion independence
* Capacity and willingness to adhere to study visit schedule and specific protocol procedures.
* Compliance with effective contraception without interruption, according to physician's judgement, from 28 days before treatment start up to at least 6 months after treatment discontinuation, agreeing not to donate semen/eggs during treatment and for at least 6 months after last treatment dose.

Exclusion Criteria:

* More than one prior systemic therapy for HL.
* Presence of autoimmune disease (based on medical history): systemic lupus erythematosus, autoimmune thyroid disease (Hashimoto's thyroiditis, Basedow's disease), Sjögren's syndrome, glomerulonephritis, multiple sclerosis, rheumatoid arthritis, vasculitis, idiopathic pulmonary fibrosis (includine bronchiolitis obliterans organizing pneumonia) and inflammatory bowel disease (Crohn's disease, ulcerative colitis).
* Previous skin toxicity (i.e. Steven-Johnson Sdr, severe skin reactions.
* Prior allogeneic stem cell transplantation or prior solid organ transplant.
* History of active tubercolosis.
* History of leptomeningeal disease.
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment.
* Central nervous system (CNS) involvement by lymphoma.
* Major surgery (excluding any lymph node biopsy) within 28 days prior to signing informed consent.
* Seropositivity for HBV or evidence of active infection. The following categories may be considered for the study:

  * HBsAg positive with HBV DNA < 2000 UI/ml (inactive carriers); HBV DNA > 2000 UI/ml is criteria of exclusion
  * HBsAg negative but HBsAb positive
  * HBsAg negative but HBcAb positive HBsAg positive with HBV DNA < 2000 UI/ml and HBsAg negative but HBcAb positive will be eligible for the study only if they accept to receive antiviral prophylaxis for all the period of treatment and at least for 12 months after the end of therapy. Treatment should be stopped in case of hepatitis reactivation. - Seropositivity for HCV. Patients with presence of HCV antibody are eligible only if PCR result are negative for HCV RNA
* Seropositivity for HIV.
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail bed) or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics except if for tumor fever) within 2 weeks of the start of Cycle 1.
* Life expectancy lower than 6 months.
* Prior history of malignancies, other than HL, unless the patient has been free for at least 5 years (exceptions: localized non-melanoma skin cancer ad carcinoma in situ of the cervix).
* Any of the following laboratory abnormalities: liver enzymes (AST/SGOT and/or ALT/SGPT) > 3 fold the upper limit of normal (except of liver involvement by lymphoma); total bilirubin > 1.5 mg/dL (except for patients with known Gilbert's disease or biliary tree compression by lymphoma masses); creatinine clearance < 30 mL/min.
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Pregnancy or breastfeeding, or unwillingness to comply with adequate contraception (one negative pregnancy test within 14 days prior to initiation of study treatment required).
* Any serious medical condition, laboratory abnormality or psychiatric illness that would prevent the patient from signing the informed consent or which may place the patient at unacceptable risk if participating in the study.

Exception to Exclusion:

* Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
* Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
* Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

  * Rash must cover < 10% of body surface area
  * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
  * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease (COPD) exacerbation) are eligible for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2027-04-27 (Estimated); Study Completion 2030-04-27 (Estimated)

PRIMARY OUTCOMES:
For Phase I part: evaluation of the maximum tolerated dose (MTD) of the atezolizumab. | During first cycle of treatment based on atezolizumab in combination with BEGEV in phase I study. Maximum time frame 17 months.
  The maximum tolerated dose (MTD) of the atezolizumab in combination with BEGEV will be established in the first cycle of therapy, in order to determine the recommended phase II dose (RP2D). Patients will be accrued in 3 patients cohorts at each dose level, starting from level 1. Dose de-escalation will be performed following the standard 3+3 rule, registering any Dose Limiting Toxicity (DLT).
For Phase II part: evaluation of the Complete Response Rate (CRR) before ASCT. | From initial treatment based on Atezolizumab and BEGEV to intensification treatment with ASCT. Time frame 4 months.
  The assessment of CRR before ASCT will be performed by an independent radiologic review committee (IRRC) according to the Lugano classification response criteria (2014) and the LYmphoma Response to Immunomodulatory Therapy Criteria (LYRIC 2016).
  CRR will be defined as the proportion of patients in CR after the first 4 cycles of induction treatment, according to Lugano classification response Criteria and LYRIC 2016 criteria. Patients without response assessment (due to whatever reason) will be considered as non-responders.

SECONDARY OUTCOMES:
For Phase II part: evaluation of the overall response rate (ORR), partial response (PR), stable disease (SD) and progression disease (PD) rates. | The best response between the date of beginning of therapy and the last restaging. Time frame 14 months.
  The assessment of the overall response rate (ORR), partial response (PR), stable disease (SD) and progression disease (PD) rates will be performed according to the Lugano 2014 criteria and LYRIC 2016 criteria.
For Phase II part: evaluation of the rate of partial response (PR) converted to Complete Response (CR). | At the end of consolidation treatment with atezolizumab in the experimental arm. Time Frame 14 months.
  The rate of PR converted to CR will be assessed as the number of PR converted in CR at the end of consolidation treatment with atezolizumab in the experimental arm.
For Phase II part: evaluation of the peripheral blood stem-cell mobilization | At the end of treatment based on atezolizumab and BEGEV. Time Frame 3 months.
  The peripheral blood stem-cell mobilization will be assessed in patients receiving atezolizumab combined to BEGEV schedule. Adequate stem cells mobilization will be defined by the target cell harvesting of 3 x 1.000.000 CD34+ cells/kg.
For Phase II part: evaluation of engraftment after ASCT | Between 30 and 60 days after ASCT: Time Frame 5 months.
  Engraftment will be assessed in patients who received ASCT after salvage treatment with atezolizumab combined to BEGEV. Engraftment will be defined as the first of three consecutive days of achieving a sustained peripheral blood neutrophil count of >500 × 1.000.000/L. Platelet engraftment is usually defined as independence from platelet transfusion for at least 7 days with a platelet count of more than >20 × 1.000.000.000/L.
For Phase II part: evaluation of duration of response (DoR). | From the CR to the date of relapse or progression or last scheduled visit. Time frame 50 months.
  The duration of response will be defined as the time from date of documented tumor response (CR) until lymphoma relapse or progression.
For Phase II part: evaluation of Progression Free Survival (PFS) for all patients. | From beginning therapy to progression or relapse disease or death. Time frame 50 months.
  PFS will be assessed for all patients and it will be defined as the time from beginning of therapy until lymphoma relapse or progression or death as a result of any cause; responding patients and patients who are lost to follow up will be censored at their last assessment date. It will be measured also in long-tem follow up in order to better assess patients' prognosis.
For Phase II part: evaluation of OS. | From the beginning of therapy to death for any cause or last scheduled visit. Time frame 50 months.
  OS will be assessed for all patients and it will be defined as the time from beginning of therapy until death as a result of any cause; alive patients and those who are lost to follow up will be censored at their last assessment date. it will be measured also in long-tem follow up in order to better assess patients' prognosis.
For Phase II part: evaluation of safety and tolerability of atezolizumab and BEGEV. | From the beginning of treatment to death or lost to follow-up or last scheduled visit. Time frame 50 months.
  The safety and the tolerability of a first salvage treatment based on the combination of intravenous (IV) atezolizumab and BEGEV regimen will be assessed throughout the study by the measurement of: patients' withdrawal rate, incidence, type and grade of any adverse event (AE) and serious adverse event (SAE) assessed by CTCAE v.4.0, hospitalization rate (except it for study therapy administration).
For Phase II part: evaluation of he correlation of quantitative baseline PET parameters | From the beginning of treatment to death or lost to follow-up or last scheduled visit. Time frame 50 months.
  To evaluate the correlation of quantitative baseline PET parameters with progression/failure free survival and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — U.O. Ematologia - Istituto Clinico Humanitas - Rozzano - ITALY
Locations (32):
- Italy (32):
  - S.C. Ematologia - A.O. SS. Antonio e Biagio e Cesare Arrigo, Alessandria, Alessandria
  - Ematologia - Fondazione del Piemonte per l'Oncologia - IRCCS, Candiolo, Turin
  - S.C. Ematologia e Trapianto emopoietico - Azienda Ospedaliera S.Giuseppe Moscati, Avellino
  - Divisione di Oncologia e dei Tumori immuto-correlati - IRCCS Centro di Riferimento Oncologico di Aviano, Aviano
  - U.O.C Ematologia - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - Ematologia - Ospedale "Monsignor Raffaele Dimiccoli", Barletta
  - Ematologia - ASST Spedali Civili di Brescia, Brescia
  - Ospedale S. Maria Goretti - UOC Ematologia con Trapianto, Latina
  - Ematologia - Ospedale Vito Fazzi, Lecce
  - IRCCS Istituto Romagnolo per lo studio dei Tumori "Dino Amadori" - IRST S.R.L. - Ematologia, Meldola
  - Azienda Ospedali Riuniti Papardo-Piemonte - S.C. Ematologia, Messina
  - Ematologia - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan
  - SC Ematologia - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto Nazionale Tumori - IRCCS Fondazione G. Pascale - UOC Ematologia Oncologica, Napoli
  - U.O. Onco-ematologia - Presidio ospedaliero "A. TORTORA", Pagani
  - Divisione di Ematologia - A.O. Ospedali Riuniti Villa Sofia-Cervello, Palermo
  - Div. di Ematologia - IRCCS Policlinico S. Matteo di Pavia, Pavia
  - Ematologia - Ospedale S. Maria della Misericordia, Perugia
  - Azienda USL Piacenza - UOC Ematologia e Centro Trapianti, Piacenza
  - Ospedale delle Croci - Ematologia, Ravenna
  - Ematologia - Azienda Unitа Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Ospedale degli Infermi di Rimini - U.O. di Ematologia, Rimini
  - Ematologia - Ospedale S. Camillo, Roma
  - Istituto Ematologia -Dipartimento di Medicina Traslazionale e di Precisione - Policlinico Umberto I - Università "La Sapienza", Roma
  - Policlinico Universitario Campus Bio-Medico - Ematologia - Trapianto cellule staminali - Medicina Trasfusionale e Terapia cellulare, Roma
  - Universitа Cattolica S. Cuore - Ematologia, Roma
  - U.O. Ematologia - Istituto Clinico Humanitas, Rozzano
  - S.C. Oncoematologia - A.O. S. Maria di Terni, Terni
  - A.O.U. Citta della Salute e della Scienza di Torino - Ematologia Universitaria, Torino
  - S.C.Ematologia - A.O.U. Città della Salute e della Scienza di Torino, Torino
  - A.O. C. Panico - U.O.C Ematologia e Trapianto, Tricase
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASUGI) - SC Ematologia, Trieste

IPD SHARING:
Plan to Share IPD: No